CLINICAL TRIAL: NCT00998335
Title: Effect of a Basal/Pre-Meal Insulin Strategy (Detemir/Aspart) to Improve Insulin Secretion and Action in Subjects With Type 2 Diabetes
Brief Title: Effect of a Basal/Pre-Meal Insulin Strategy (Detemir/Aspart) on Insulin Secretion and Action in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20060167
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes mellitus; Insulin therapy; Detemir (Levemir); Aspart (Novolog); Hepatic steatosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Fatty Liver | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin detemir only (Active Comparator): Patients with uncontrolled T2DM are treated with insulin detemir for 6 months. Insulin detemir is given at bedtime aiming at a fasting plasma glucose between 80-100 mg/dl. This group will receive Long-acting bedtime insulin detemir (Levemir).
  Interventions: Drug: Long-acting bedtime insulin detemir (Levemir)
- Insulin detemir plus aspart (Experimental): After baseline evaluations, insulin detemir will be given at bedtime and titrated to achieve a fasting plasma glucose between 80-100 mg/dl. After 3 months patients will be admitted to assess the metabolic effects of intervention. After this, insulin aspart (insulin detemir plus aspart) will be added before breakfast, lunch and dinner titrated to normalize the postprandial plasma glucose. After another 3 months patients are readmitted and all study procedures repeated. This group will receive Insulin detemir and pre-meal insulin aspart.
  Interventions: Drug: Insulin detemir and pre-meal insulin aspart.

INTERVENTIONS:
Drug: Long-acting bedtime insulin detemir (Levemir) — This group will receive Insulin detemir. Insulin detemir is given at bedtime aiming at a fasting plasma glucose between 80-100 mg/dl.
  Other Names: Levemir insulin (trademark insulin by Novo Nordisk)
  Arms: Insulin detemir only
Drug: Insulin detemir and pre-meal insulin aspart. — This group will receive Insulin detemir plus aspart. The group will start with Insulin detemir at bedtime. Then in three months they will Insulin aspart before breakfast, lunch and dinner.
  Other Names: Insulin detemir = Levemir (Novo Nordisk); Insulin aspart = Novolog (Novo Nordisk)
  Arms: Insulin detemir plus aspart

SUMMARY:
The optimal insulin therapy in T2DM is controversial and its impact on nonalcoholic fatty liver disease (NAFLD) has not been systematically studied before, and in particular, never when using the new insulin formulations detemir (Levemir®) or aspart (Novolog®). This study is to determine the effect on hepatic steatosis and insulin secretion/action of lowering the fasting plasma glucose (FPG) to target with once daily basal insulin detemir alone or combining insulin detemir with premeal insulin aspart in patients with uncontrolled type 2 diabetes mellitus (T2DM).

In the first 3 months the investigators will optimize metabolic control in all patients with intensive basal (bedtime) detemir insulin aiming at a normal fasting plasma glucose. After this treatment period, patients will be randomized in the second 3 months in a 2:1 ratio to insulin detemir or detemir plus aspart. The investigators propose that insulin will improve day-long glycemic control and A1c, reduce hepatic steatosis (NAFLD) (primary endpoint) and insulin secretion/sensitivity being well tolerated while causing minimal weight gain and hypoglycemia (secondary endpoints). The study will allow to assess if there is an additional benefit of adding pre-meal rapid-acting insulin aspart to basal insulin to these endpoints.

DETAILED DESCRIPTION:
The control of hyperglycemia in T2DM ameliorates the metabolic abnormalities of T2DM but whether this improves hepatic steatosis has not been examined carefully with the use of improved insulin formulations (long-acting insulins detemir or glargine, alone or combined with pre-meal short-acting insulins). Most research studies have focused on glycemic control without a careful examination to the underlying mechanisms, with some of these studies reporting on improved hepatic and muscle insulin sensitivity. The investigators have found in the laboratory that intensified insulin therapy in T2DM is associated with enhanced glycogen synthase fractional velocity and non-oxidative glucose disposal, but with no improvement at the level of insulin-stimulated insulin receptor tyrosine phosphorylation, hexokinase II mRNA or enzyme function, phosphatidylinositol 3-kinase (PI 3-kinase) associated with IRS-1, or Akt phosphorylation. Our work did not examine hepatic steatosis or insulin secretion/action, nor was designed to distinguish between the relative contribution of reduced glucotoxicity on insulin sensitivity vs. beta-cell function from pre-meal regular vs. NPH insulin. It is possible that the beneficial effects of insulin therapy of reduced plasma glucose and FFA concentrations may be offset by excessive hyperinsulinemia and weight gain from the use of insulins with suboptimal pharmacokinetics compared to the newer insulin formulations.

Insulin detemir is an insulin analogue approved in 2005 by the FDA. It is a long-acting insulin analogue that has shown to be more predictable in achieving therapeutic plasma insulin levels compared to NPH insulin. This is associated with several clinical benefits, such as better glycemic control, less hypoglycemia, modest weight gain and better quality of life for patients with type 2 diabetes. If gluco-lipotoxicity likely play an important role in the development of hepatic steatosis (NAFLD) in T2DM the investigators speculate that if reversed by a strategy of basal long-acting insulin (insulin detemir) alone, or combined with a rapid-acting analog (pre-meal insulin aspart) may be a good strategy for the treatment of T2DM.

ELIGIBILITY:
Inclusion Criteria:

To participate patients must:

1. Be able to communicate meaningfully with the Investigator and be legally competent to provide written informed consent.
2. Female patients must be non-lactating and must either be at least two years post-menopausal, or be using adequate contraceptive precautions (i.e. oral contraceptives, approved hormonal implant, intrauterine device, diaphragm with spermicide, condom with spermicide), or be surgically sterilized (i.e. bilateral tubal ligation, bilateral oophorectomy). Female patients who have undergone a hysterectomy are eligible for participation in the study. Female patients (except for those patients who have undergone a hysterectomy or a bilateral oophorectomy) are eligible only if they have a negative pregnancy test throughout the study period.
3. Age range of 18 to 70 years (inclusive).
4. Patients must have been on a stable dose of allowed chronic medications for two months prior to entering the double-blind treatment period.
5. All participants must have the following laboratory values:

   * Hemoglobin ≥ 12 g/dl in males or ≥ 11 g/dl in females
   * Serum creatinine ≤ 1.5 mg/dl
   * AST (SGOT) ≤ 2.5 times upper limit of normal
   * ALT (SGPT) ≤ 2.5 times upper limit of normal
   * Alkaline phosphatase ≤ 2.5 times upper limit of normal

Exclusion Criteria:

Patients will be excluded if any of the following criteria are present:

1. Individuals with type 1 diabetes or type 2 diabetes and a FPG ≥ 300 mg/dl.
2. Subjects on sulfonylureas, metformin and/or TZDs unless the dose has been stable for at least 2 months prior to study entry.
3. Patients on any of the following medications: thiazide or furosemide diuretics, beta-blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless the patient has been on stable doses of such agents for the past two months before entry into the study. Patients may be taking stable doses of estrogens or other hormonal replacement therapy if the patient has been on these agents for the prior two months. Patients taking systemic glucocorticoids will be excluded.
4. Past (within 1 year) or current history of alcohol abuse.
5. Patients will be excluded if there is a history of clinically significant heart disease (New York Heart Classification greater than grade II), peripheral vascular disease (history of claudication), or pulmonary disease (dyspnea on exertion of one flight or less; abnormal breath sounds on auscultation) or chronic renal failure (serum creatinine greater than 1.5 mg/dl).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cusi, M.D., Principal Investigator — University of Flordia
Locations (1):
- The University of Texas H.S.C. at San Antonio and the San Antonio Audie L. Murphy VA Hospital, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical Research Unit
Pre-assignment Details: All participants started in the "Insulin detemir only" arm. At week 12 the participants were randomized in a 2:1 ratio to either Insulin detemir only arm or to Insulin detemir plus aspart.
Groups:
- Insulin Detemir Only: Patients with uncontrolled T2DM are treated with insulin detemir for 6 months
  Long-acting bedtime insulin detemir (Levemir) : Insulin detemir is given at bedtime aiming at a fasting plasma glucose between 80-100 mg/dl.
- Insulin Detemir Plus Aspart: After baseline evaluations (admission #1) insulin detemir will be given at bedtime and titrated to achieve a fasting plasma glucose between 80-100 mg/dl. After 3 months patients will be admitted to assess the metabolic effects of intervention. After this, insulin aspart will be added before breakfast, lunch and dinner titrated to normalize the postprandial plasma glucose. After another 3 months patients are readmitted and all study procedures repeated as during admissions #1 and #2.
  Insulin detemir and pre-meal insulin aspart. : Insulin detemir at bedtime. Insulin aspart before breakfast, lunch and dinner.
Period: Initial Treatment (Months 0 - 3)
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Started | 30 | 0
Completed | 30 | 0
Not Completed | 0 | 0
Period: Randomized Period (Months 3 to 6)
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Started | 8 (All participants started in the "Insulin detemir only" arm. At month 3 subjects were randomized 2:1.) | 22 (All participants started in the "Insulin detemir only" arm. At month 3 subjects were randomized 2:1.)
Completed | 8 | 20
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants were started in the "Insulin detemir only" arm. At week 12 the participants were randomized in a 2:1 ratio between the two arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart | Total
Number analyzed (Participants) | 8 | 22 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 22 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (8) | 59 (8) | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 8 | 19 | 27
Region of Enrollment [Number; unit: participants]
  United States | 8 | 22 | 30

OUTCOME MEASURES:

1. Primary Outcome: Hepatic Steatosis
Description: Hepatic steatosis measured by proton magnetic resonance spectroscopy (1H-MRS).
Time Frame: 3 and 6 months
Population: In six patients liver MRS was not possible due to claustrophobia, metal parts, or too large for MRI scanner. N=30 participants in the Insulin detemir x 3 months, N=8 participants in the Insulin Detemir alone and 22 in the Detemir Plus Aspart at 6 months.
Measure: Mean (Standard Deviation); unit: percentage of liver fat
Groups:
- Insulin Detemir x 3 Months (All Pts Had Liver MRS): Liver fat by MRS measured after 3 months of insulin.
Arm/Group | Insulin Detemir x 3 Months (All Pts Had Liver MRS) | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
percentage of liver fat
  Month 3 | 6.7 (4.4) | NA (NA) — Participants were only randomized to this arm after 3 months of treatment.
  Month 6 | 8.4 (7.2) | 5.9 (4.2)
Statistical Analysis 1: Comparison: Insulin Detemir x 3 Months (All Pts Had Liver MRS); Baseline versus 3 months; Test type: Superiority or Other; p = 0.03, ANOVA

2. Secondary Outcome: Metabolic Control as Measured by the A1c
Time Frame: 3 and 6 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: percentage of A1c
Groups:
- Insulin Detemir Only (3 and 6 Months): All patients with uncontrolled T2DM are treated with insulin detemir for 6 months and after 3 months randomized to either arm. Long-acting bedtime insulin detemir (Levemir) : Insulin detemir is given at bedtime aiming at a fasting plasma glucose between 80-100 mg/dl.
Arm/Group | Insulin Detemir Only (3 and 6 Months) | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
percentage of A1c
  3-month - A1c | 7.4 (1.4) | NA (NA) — Participants were not randomized into this arm until month 3.
  6-month - A1c | 6.9 (0.5) | 6.7 (0.7)

3. Secondary Outcome: Change in Insulin Secretion
Description: Derived from the hyperglycemic clamp (Plasma C-peptide change vs. pretreatment in first and second phase).
Time Frame: 3 and 6 months.
Population: All participants were started in the "Insulin detemir only" arm. At week 12 the participants were randomized in a 2:1 ratio between the two arms. N=30 at 3 months and N=28 at 6 months.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Insulin Detemir Only (3 and 6 Months): All patients with uncontrolled T2DM are treated with insulin detemir for 6 months and after 3 months randomized to either arm. Long-acting bedtime insulin detemir (Levemir) is given at bedtime aiming at a fasting plasma glucose between 80-100 mg/dl.
Arm/Group | Insulin Detemir Only (3 and 6 Months) | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
ng/ml
  3-month C-peptide level increase in first phase | 0.5 (1.3) | NA (NA) — Participants were not randomized to this arm until month 3.
  3-month C-peptide level increase in second phase | 1.6 (2.5) | NA (NA) — Participants were not randomized to this arm until month 3.
  6-month C-peptide level increase in first phase | -0.1 (0.9) | 0.2 (1.4)
  6-month C-peptide level increase in second phase | 0.6 (2.0) | 0.2 (2.3)

4. Secondary Outcome: Intramyocellular (IMCL) by Magnetic Resonance Imaging and Spectroscopy (MRS).
Description: Percent intramyocellular (IMCL) by magnetic resonance imaging and spectroscopy (MRS).
Time Frame: 3 and 6 months.
Population: All participants were started in the "Insulin detemir only" arm. At week 12 the participants were randomized in a 2:1 ratio between the two arms. N=30 for first 3 months and N=28 for 6 months
Measure: Mean (Standard Deviation); unit: % of intramyocellular triglyceride
Groups:
- Insulin Detemir Only: Patients with uncontrolled T2DM are treated with insulin detemir for 6 months. After patients were treated for 3 months with bedtime insulin detemir they were randomized to either continue with bedtime insulin detemir or add premeal rapid-acting insulin novolog.
  Long-acting bedtime insulin detemir (Levemir) was given at bedtime aiming at a fasting plasma glucose between 80-100 mg/dl.
- Insulin Detemir Plus Aspart: After baseline evaluations (admission #1) insulin detemir will be given at bedtime and titrated to achieve a fasting plasma glucose between 80-100 mg/dl. After 3 months patients will be admitted to assess the metabolic effects of intervention. After this, insulin aspart will be added before breakfast, lunch and dinner titrated to normalize the postprandial plasma glucose. After another 3 months patients are readmitted and all study procedures repeated as during admissions #1 and #2.
  Insulin detemir was given at bedtime. Insulin aspart before breakfast, lunch and dinner.
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
% of intramyocellular triglyceride
  3-month intramyocellular triglycerides | 0.63 (0.62) | NA (NA) — Participants were not randomized to this arm until month 3.
  6-month intramyocellular triglycerides | 1.05 (0.18) | 0.49 (0.47)

5. Secondary Outcome: Plasma Lipid Concentration.
Description: Fasting plasma lipid concentration on day of admission at 3 and 6 months.
Time Frame: 3 and 6 months.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
mg/dL
  3-month total cholesterol | 136 (36) | NA (NA) — Participants were not randomized to this arm until month 3.
  3-month LDL-cholesterol | 76 (27) | NA (NA) — Participants were not randomized to this arm until month 3.
  3-month triglycerides | 154 (76) | NA (NA) — Participants were not randomized to this arm until month 3.
  3-month HDL-C | 33 (8) | NA (NA) — Participants were not randomized to this arm until month 3.
  6-month total cholesterol | 147 (31) | 145 (37)
  6-month LDL-cholesterol | 86 (29) | 80 (28)
  6-month triglycerides | 150 (66) | 144 (62)
  6-month HDL-C | 31 (5) | 33 (7)

6. Secondary Outcome: Change in Anthropometric Measure (Body Weight).
Description: Change in anthropometric measure (body weight) done on day of admission at 3 and 6 months.
Time Frame: 3 and 6 months.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Change from baseline (Kg)
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
Change from baseline (Kg)
  3-month total body weight | -0.8 (7.3) | NA (NA) — Participants were not randomized to this arm until month 3.
  6-month total body weight | 0.8 (1.9) | 0.3 (3.5)

7. Secondary Outcome: Number of Hypoglycemic Events
Description: Defined as hypoglycemia <40 mg/dl and/or requiring medical assistance during the trial.
Time Frame: 3 and 6 months
Population: as for outcome 4
Measure: Number; unit: Number of events
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
Number of events
  3-month rate of severe hypoglycemia | 0 | NA — Participants were not randomized to this arm until month 3.
  6-month rate of severe hypoglycemia | 0 | 0

8. Secondary Outcome: Metabolic Control as Measured by the Fasting Plasma Glucose Concentration
Time Frame: 3 and 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir Only (3 and 6 Months) | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
mg/dL
  3-month - Fasting plasma glucose | 105 (38) | NA (NA) — Participants were not randomized to this arm until month 3.
  6-month - Fasting plasma glucose | 89 (18) | 116 (27)

9. Secondary Outcome: Metabolic Control as Measured by the Postprandial Plasma Glucose During the Day-long Plasma Glucose Profile.
Time Frame: 3 and 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Detemir Only (3 and 6 Months) | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
mg/dL
  3-month - Day-long plasma glucose profile | 168 (44) | NA (NA) — Participants were not randomized until month 3
  6-month - Day-long plasma glucose profile | 153 (38) | 170 (48)

10. Secondary Outcome: Advanced Lipid Testing
Description: Change in lipoprotein particle number was determined using NMR.
Time Frame: 3 and 6 months
Measure: Mean (Standard Deviation); unit: Change in number of particles (nmol/L)
Arm/Group | Insulin Detemir Only (3 and 6 Months) | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
Change in number of particles (nmol/L)
  VLDL particles (3 months) | -15 (39) | NA (NA) — Randomization of this group occurred at month 3.
  VLDL particles (6 months) | -5 (38) | -2 (31)
  LDL particles (3 months) | -100 (313) | NA (NA) — Randomization of this group occurred at month 3.
  LDL particles (6 months) | 128 (206) | 85 (209)
  HDL particles (3 months) | 0 (3) | NA (NA) — Randomization of this group occurred at month 3.
  HDL particles (6 months) | 2 (4) | 1 (4)

11. Secondary Outcome: Change in Anthropometric Measure (Body Mass Index [BMI]).
Description: Change in anthropometric measure (body mass index [BMI]) done on day of admission at 3 and 6 months.
Time Frame: 3 and 6 months.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Change from baseline (Kg/m2)
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
Change from baseline (Kg/m2)
  3-month body mass index | -0.4 (2.7) | NA (NA) — Patients were not randomized to this arm until month 3.
  6-month body mass index | 0.3 (0.6) | 0.2 (1.2)

12. Secondary Outcome: Percent Change From Baseline in Vascular Inflammatory Markers
Description: Inflammatory Markers include: Adiponectin, MMP-9, E-selectin, sICAM, and sVCAM
Time Frame: 3 and 6 months
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Number analyzed (Participants) | 30 | 22
Percentage of change
  Adiponectin (3 months) | 18 (63) | NA (NA) — Patients were not randomized to this arm until month 3.
  Adiponectin (6 months) | 65 (71) | 5 (30)
  MMP-9 (3 months) | 32 (59) | NA (NA) — Patients were not randomized to this arm until month 3.
  MMP-9 (6 months) | 30 (115) | 49 (73)
  E-selectin (3 months) | -6 (25) | NA (NA) — Patients were not randomized to this arm until month 3.
  E-selectin (6 months) | 34 (34) | 19 (29)
  sICAM (3 months) | -4 (22) | NA (NA) — Patients were not randomized to this arm until month 3.
  sICAM (6 months) | 2 (12) | -1 (15)
  sVCAM (3 months) | 1 (8) | NA (NA) — Patients were not randomized to this arm until month 3.
  sVCAM (6 months) | 14 (13) | 7 (11)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Insulin Detemir Only | Insulin Detemir Plus Aspart
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/22
Other Adverse Events (participants affected / at risk) | 0/30 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No